CLINICAL TRIAL: NCT00575874
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose and Active Comparator-Controlled Dose-Response Study of Rivoglitazone (CS-011) in Patients With Type 2 Diabetes
Brief Title: Placebo and Active Comparator Controlled Dose Response Study of Rivoglitazone in Type 2 Diabetes
Acronym: RAISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Dr. Alice Pik Shan Kong, The Chinese University of Hong Kong
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS011-A-J205
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes
Keywords: rivoglitazone HCl; pioglitazone HCl; thiazolidinedione; peroxisome proliferator-activated receptor gamma (PPAR gamma); type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 0.5 mg rivoglitazone HCl tablets once daily for 12 weeks
  Interventions: Drug: Rivoglitazone HCl
- 2 (Experimental): 1.0 mg rivoglitazone HCl tablets once daily for 12 weeks
  Interventions: Drug: rivoglitazone HCl
- 3 (Experimental): 1.5 mg rivoglitazone HCl tablets once daily for 12 weeks
  Interventions: Drug: rivoglitazone HCl
- 4 (Active Comparator): 30 mg pioglitazone HCl capsules once daily for 12 weeks
  Interventions: Drug: pioglitazone HCl
- 5 (Placebo Comparator): Matching rivoglitazone HCL placebo tablets and/or matching pioglitazone HCL placebo capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rivoglitazone HCl — 0.5 mg rivoglitazone HCl tablets once daily for 12 weeks
  Arms: 1
Drug: rivoglitazone HCl — 1.0 mg rivoglitazone HCl tablets once daily for 12 weeks
  Arms: 2
Drug: rivoglitazone HCl — 1.5 mg rivoglitazone HCl tablets once daily for 12 weeks
  Arms: 3
Drug: pioglitazone HCl — 30 mg capsules once daily for 12 weeks
  Arms: 4
Drug: placebo — matching tablets or capsule once daily for 12 weeks
  Arms: 5

SUMMARY:
The purpose of the study is to assess the efficacy response of rivoglitazone HCl compared to pioglitazone HCl on the placebo-corrected change from baseline in HbA1c after 12 weeks of treatment in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* HbA1c >6.5% and <10.0%
* FPG >126 mg/dL (7 mmol/L) and < 270 mg/dL (15 mmol/L)

Exclusion Criteria:

* History of type 1 diabetes
* History of ketoacidosis
* Current insulin therapy
* C-peptide <0.5ng/mL
* Imparied hepatic function
* NYHA Class II-IV cardiac status or hospitalization for CHF or EF<40%
* uncontrolled hypertension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline for rivoglitazone HCl compared to that for placebo | 12 weeks

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose from baseline for rivoglitazone HCl compared to that for placebo. Change in HbA1c from baseline compared to that for pioglitazone HCl | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong, China